CLINICAL TRIAL: NCT01913522
Title: Cryoballoon vs. Irrigated Radiofrequency Catheter Ablation: The Effect of Double Short vs. Standard Exposure Cryoablation Duration During Pulmonary Vein Isolation.
Brief Title: Cryoballoon vs. Irrigated Radiofrequency Catheter Ablation: Double Short vs. Standard Exposure Duration
Acronym: CIRCA-DOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jason Andrade, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H13-01689
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard cryoablation (Experimental): Patients randomized to the standard group will undergo cryoablation with target duration of 240 seconds. Once PVI is achieved a single "bonus" application of 240 seconds will be delivered after the rewarming phase (to +20oC).
  Interventions: Procedure: Pulmonary Vein Isolation
- Irrigated RF Ablation (Active Comparator): Patients randomized to irrigated RF group will undergo standard wide circumferential PVI with an irrigated radiofrequency catheter
  Interventions: Procedure: Pulmonary Vein Isolation
- Short Cryoablation (Experimental): Patients randomized to the multiple-freeze group will undergo cryoablation with target duration of 120 seconds. Once PVI is achieved a single "bonus" application of 120 seconds will be delivered after the rewarming phase (to +20oC).
  Interventions: Procedure: Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia and is associated with reductions in quality of life, functional status, cardiac performance, and overall survival.1 Catheter ablation, which is centered on electrical isolation of triggering foci within the pulmonary veins (PVI) through circumferential lesions around PV ostia, has been shown to result in sustained improvements in quality of life, decreased hospitalizations and, potentially, improved survival.2-4 PVI can be accomplished by percutaneous catheter-based thermo-coagulation (burning) with radiofrequency (RF) energy delivery or alternatively by thermo-cooling (freezing) with a cryoballoon catheter.5 Cryothermal ablation with a cryoballoon catheter offers an efficacious means to achieve PVI that is safer than the established technique. Although cryoballoon ablation has been used in clinical practice for sometime, the optimal duration of cryoballoon ablation has not been determined. Moreover, the biophysics of cryo-lesion formation suggests that repeated short freezes ("freeze-thaw-freeze" cycles) may be more efficacious in achieving deep homogenous lesion when compared to prolonged freezing durations. This grant proposal is to verify if repeated short freezing cycles are more efficacious (i.e., fewer recurrence of AF), and safer, than the established standard of long, single freeze cycles.

ELIGIBILITY:
Inclusion Criteria:

- Non-permanent atrial fibrillation documented on a 12 lead ECG, TTM or Holter monitor within the last 12 months Low Burden Paroxysmal - ≥2 episodes of AF over the past 12 months; Episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.

High Burden Paroxysmal - ≥4 episodes of AF over the past 6 months, with ≥2 episodes >6 hours in duration; Episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.

Early Persistent - ≥2 episodes of AF over the past 12 months; Episodes are successfully terminated via cardioversion within 7 days of onset.

* Age of 18 years or older on the date of consent
* Candidate for ablation based on AF that is symptomatic and refractory (ineffective or intolerant) to at least one class 1 or 3 antiarrhythmic
* Continuous anticoagulation with warfarin (INR 2-3), low molecular weight heparin, or a novel oral antithrombotic (dabigatran, apixaban, rivaroxaban) for ≥4 weeks prior to the ablation; or a TEE that excludes LA thrombus ≤48 hours before ablation
* Informed Consent Form

Exclusion Criteria:

* Previous left atrial (LA) ablation or LA surgery
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Anteroposterior LA diameter greater than 5.5 cm by TTE
* Cardiac valve prosthesis
* Clinically significant (moderately-severe, or severe) mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* NYHA class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) less than 35%
* Hypertrophic cardiomyopathy
* Significant CKD (eGFR <30 mL/min/m2)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (strokes or TIAs) during the six-month interval preceding the consent date
* Subject known to be pregnant
* Life expectancy less than one (1) year
* Currently participating or anticipated to participate in any other clinical trial of a drug, device or biologic during the duration of this study
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence of AF, atrial flutter, or left atrial tachycardia documented by 12-lead ECG, surface ECG rhythm strips, ambulatory ECG monitor, or implantable loop recorder and lasting 30 seconds or longer | 1 year

SECONDARY OUTCOMES:
Time to first recurrence of symptomatic electrocardiographically documented AF/AFL/AT between days 91 and 365 after ablation | 1 year
Total arrhythmia burden (daily AF burden - hours/day; overall AF burden - % time in AF) | 1 year
Repeat ablation procedure because of documented recurrence of symptomatic AF/AFL/AT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason Andrade, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Aguilar M, Macle L, Honfo SH, Khairy P, Cadrin-Tourigny J, Sidhu A, Deyell MW, Hawkins NM, Bennett RG, Andrade JG. Blanking Period After Catheter Ablation of Paroxysmal Atrial Fibrillation: Insights From Continuous Cardiac Monitoring. Circ Arrhythm Electrophysiol. 2025 Mar;18(3):e013232. doi: 10.1161/CIRCEP.124.013232. Epub 2025 Feb 18. No abstract available. PMID 39963799
- [Derived] Andrade JG, Bennett RG, Deyell MW, Bennett MT, Phulka J, Hawkins NM, Aksu T, Field TS, Aguilar M, Khairy P, Macle L. Long-Term Differences in Autonomic Alterations After Cryoballoon vs Radiofrequency Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2025 Jan;11(1):19-29. doi: 10.1016/j.jacep.2024.09.003. Epub 2024 Oct 30. PMID 39480391
- [Derived] Aguilar M, Macle L, Deyell MW, Yao R, Hawkins NM, Khairy P, Andrade JG. Influence of Monitoring Strategy on Assessment of Ablation Success and Postablation Atrial Fibrillation Burden Assessment: Implications for Practice and Clinical Trial Design. Circulation. 2022 Jan 4;145(1):21-30. doi: 10.1161/CIRCULATIONAHA.121.056109. Epub 2021 Nov 24. PMID 34816727
- [Derived] Samuel M, Khairy P, Champagne J, Deyell MW, Macle L, Leong-Sit P, Novak P, Badra-Verdu M, Sapp J, Tardif JC, Andrade JG. Association of Atrial Fibrillation Burden With Health-Related Quality of Life After Atrial Fibrillation Ablation: Substudy of the Cryoballoon vs Contact-Force Atrial Fibrillation Ablation (CIRCA-DOSE) Randomized Clinical Trial. JAMA Cardiol. 2021 Nov 1;6(11):1324-1328. doi: 10.1001/jamacardio.2021.3063. PMID 34406350
- [Derived] Tang LYW, Hawkins NM, Ho K, Tam R, Deyell MW, Macle L, Verma A, Khairy P, Sheldon R, Andrade JG; CIRCA-DOSE Study Investigators. Autonomic Alterations After Pulmonary Vein Isolation in the CIRCA-DOSE (Cryoballoon vs Irrigated Radiofrequency Catheter Ablation) Study. J Am Heart Assoc. 2021 Feb;10(5):e018610. doi: 10.1161/JAHA.120.018610. Epub 2021 Feb 26. PMID 33634706
- [Derived] Yao RJR, Macle L, Deyell MW, Tang L, Hawkins NM, Sedlak T, Nault I, Verma A, Khairy P, Andrade JG; CIRCA-DOSE Study Investigators. Impact of Female Sex on Clinical Presentation and Ablation Outcomes in the CIRCA-DOSE Study. JACC Clin Electrophysiol. 2020 Aug;6(8):945-954. doi: 10.1016/j.jacep.2020.04.032. Epub 2020 Jul 29. PMID 32819529
- [Derived] Andrade JG, Macle L, Verma A, Deyell MW, Champagne J, Dubuc M, Leong-Sit P, Novak P, Roux JF, Sapp J, Khoo C, Rizkallah J, Levesque S, Tang ASL, Khairy P; CIRCA-DOSE Study Investigators. Quality of Life and Health Care Utilization in the CIRCA-DOSE Study. JACC Clin Electrophysiol. 2020 Aug;6(8):935-944. doi: 10.1016/j.jacep.2020.04.017. PMID 32819528
- [Derived] Andrade JG, Deyell MW, Verma A, Macle L, Champagne J, Leong-Sit P, Novak P, Badra-Verdu M, Sapp J, Khairy P, Nattel S. Association of Atrial Fibrillation Episode Duration With Arrhythmia Recurrence Following Ablation: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Jul 1;3(7):e208748. doi: 10.1001/jamanetworkopen.2020.8748. PMID 32614422
- [Derived] Andrade JG, Yao RRJ, Deyell MW, Hawkins NM, Rizkallah J, Jolly U, Khoo C, Raymond JM, McKinney J, Cheung C, Steinberg C, Ha A, Ramanathan K, Luong C, Glover B, Verma A, Macle L, Khairy P; CIRCA-DOSE Study Investigators. Clinical assessment of AF pattern is poorly correlated with AF burden and post ablation outcomes: A CIRCA-DOSE sub-study. J Electrocardiol. 2020 May-Jun;60:159-164. doi: 10.1016/j.jelectrocard.2020.03.008. Epub 2020 Mar 21. PMID 32371199
- [Derived] Andrade JG, Deyell MW, Nattel S, Khairy P, Dubuc M, Champagne J, Leong-Sit P, Jolly U, Badra-Verdu M, Sapp J, Verma A, Macle L; CIRCA-DOSE Study Investigators. Prevalence and clinical impact of spontaneous and adenosine-induced pulmonary vein reconduction in the Contact-Force vs. Cryoballoon Atrial Fibrillation Ablation (CIRCA-DOSE) study. Heart Rhythm. 2020 Jun;17(6):897-904. doi: 10.1016/j.hrthm.2020.01.017. Epub 2020 Jan 21. PMID 31978593
- [Derived] Andrade JG, Champagne J, Dubuc M, Deyell MW, Verma A, Macle L, Leong-Sit P, Novak P, Badra-Verdu M, Sapp J, Mangat I, Khoo C, Steinberg C, Bennett MT, Tang ASL, Khairy P; CIRCA-DOSE Study Investigators. Cryoballoon or Radiofrequency Ablation for Atrial Fibrillation Assessed by Continuous Monitoring: A Randomized Clinical Trial. Circulation. 2019 Nov 26;140(22):1779-1788. doi: 10.1161/CIRCULATIONAHA.119.042622. Epub 2019 Oct 21. PMID 31630538
- [Derived] Andrade JG, Deyell MW, Badra M, Champagne J, Dubuc M, Leong-Sit P, Macle L, Novak P, Roux JF, Sapp J, Tang A, Verma A, Wells GA, Khairy P. Randomised clinical trial of cryoballoon versus irrigated radio frequency catheter ablation for atrial fibrillation-the effect of double short versus standard exposure cryoablation duration during pulmonary vein isolation (CIRCA-DOSE): methods and rationale. BMJ Open. 2017 Oct 5;7(10):e017970. doi: 10.1136/bmjopen-2017-017970. PMID 28982836